CLINICAL TRIAL: NCT03283085
Title: A Phase 3 Long-term Safety Extension Study of SHP647 in Subjects With Moderate to Severe Ulcerative Colitis or Crohn's Disease (AIDA)
Brief Title: A Safety Extension Study of Ontamalimab in Participants With Moderate to Severe Ulcerative Colitis or Crohn's Disease (AIDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP647-304; 2017-000574-11 (EudraCT Number)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Immunosuppressants; Mesalamine; Ulcerative Colitis; Crohn's disease; Gastroenteritis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Gastroenteritis | interventions — ontamalimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Ulcerative Colitis (UC): Ontamalimab 25 mg (Experimental): Participants received 25 milligrams (mg) of ontamalimab solution for injection subcutaneously (SC), every 4 weeks (Q4W), for up to 3 years.
  Interventions: Drug: 25 mg Ontamalimab
- UC: Ontamalimab 25mg then 75 mg (Experimental): Participants received 25 mg of ontamalimab solution for injection SC, Q4W, and later progressed to receive 75 mg in a similar manner for up to 5.79 years.
  Interventions: Drug: 25 mg Ontamalimab; Drug: 75 mg Ontamalimab
- UC: Ontamalimab 75 mg (Experimental): Participants received 75 mg of ontamalimab solution for injection SC, Q4W, for up to 5.79 years.
  Interventions: Drug: 75 mg Ontamalimab
- Crohn's disease (CD): Ontamalimab 25 mg (Experimental): Participants received 25 mg of ontamalimab solution for injection SC, Q4W, for up to 3 years.
  Interventions: Drug: 25 mg Ontamalimab
- CD: Ontamalimab 25mg then 75 mg (Experimental): Participants received 25 mg of ontamalimab solution for injection SC, Q4W, and later progressed to receive 75 mg in a similar manner for up to 5.79 years.
  Interventions: Drug: 25 mg Ontamalimab; Drug: 75 mg Ontamalimab
- CD: Ontamalimab 75 mg (Experimental): Participants received 75 mg of ontamalimab solution for injection SC, Q4W, for up to 5.79 years.
  Interventions: Drug: 75 mg Ontamalimab

INTERVENTIONS:
Drug: 25 mg Ontamalimab — Ontamalimab SC solution for injection
  Other Names: PF-00547659; SHP647
  Arms: CD: Ontamalimab 25mg then 75 mg; Crohn's disease (CD): Ontamalimab 25 mg; UC: Ontamalimab 25mg then 75 mg; Ulcerative Colitis (UC): Ontamalimab 25 mg
Drug: 75 mg Ontamalimab — Ontamalimab SC solution for injection
  Other Names: SHP647; PF-00547659
  Arms: CD: Ontamalimab 25mg then 75 mg; CD: Ontamalimab 75 mg; UC: Ontamalimab 25mg then 75 mg; UC: Ontamalimab 75 mg

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of long-term treatment with ontamalimab in participants with moderate to severe Ulcerative Colitis (UC) or Crohn's disease (CD)

ELIGIBILITY:
Inclusion Criteria:

Participants with Ulcerative Colitis (UC):

* Participants and/or their parent or legally authorized representative must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Participants must be able to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent and/or assent, as applicable, to participate in the study.
* Participants must have been enrolled previously in study SHP647-301 (NCT03259334), SHP647-302 (NCT03259308), and are in the treatment period of Study SHP647-303, completed the early termination (ET) or Week 52 visit in maintenance study SHP647-303 (NCT03290781), had responded to ontamalimab treatment (in the induction and/or maintenance studies), and meet one of the following criteria:

  a. Participants are on placebo at the maintenance study ET or Week 52 visit: they received ontamalimab in the induction studies and fulfilled the maintenance study response criteria, OR b. Participants have received ontamalimab at the maintenance study ET or Week 52 visit: i) Clinical composite score that has decreased by >or=2 points and >or=30%, with an accompanying decrease in the subscore for RB >or=1 point or a subscore for RB <or=1, compared to the baseline value for induction studies, and/or ii) Composite score that has decreased by >or=30% and >or=3 points compared to the baseline value for induction studies.
* Participants receiving any treatment(s) for UC are eligible provided they have been on a stable dose for the designated period of time.

Participants with Crohn's Disease:

* Participants and/or their parent or legally authorized representative must have an understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Participants must be able to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent and/or assent, as applicable, to participate in the study.
* Participants must have been enrolled previously in Study SHP647-305 (NCT03559517) or SHP647-306 (NCT03566823) and are in the treament period of Study SHP647-307 (NCT03627091), completed the ET or Week 52 visit in maintenance study SHP647-307, had responded to ontamalimab treatment (in the induction or maintenance studies) and meet one of the following criteria:

  1. Participants are on placebo at the maintenance study ET or Week 52 visit: they received ontamalimab in the induction study and fulfilled the maintenance study response criteria, OR
  2. Participants have received ontamalimab at the maintenance study ET or Week 52 visit:

  i) CDAI score that has decreased by >or=100 points at EOT visit compared to the baseline value for induction studies, and/or ii) SES-CD that has decreased by >or=25% compared to the baseline value for induction studies.
* Participants receiving any treatment(s) for CD are eligible provided they have been on a stable dose for the designated period of time.

Exclusion Criteria:

Participants with UC:

* Participants who had major protocol deviation(s) (as determined by the sponsor) in study SHP647-301, SHP647-302, or SHP647-303.
* Participants who permanently discontinued investigational product because of an AE, regardless of relatedness to investigational product, in study SHP647-301, SHP647-302, or SHP647-303.
* Participants who are likely to require major surgery for UC.
* Participants are females who became pregnant during study SHP647-301, SHP647-302, or SHP647-303, females who are lactating, females who are planning to become pregnant during the study period, or males or females of childbearing potential not agreeing to continue using appropriate contraception methods (i.e. highly effective methods for female and medically appropriate methods for male study participants) through the conclusion of study participation.
* Participants who do not agree to postpone donation of any organ or tissue, including male participants who are planning to bank or donate sperm and female participants who are planning to harvest or donate eggs, for the duration of the study and through 16 weeks after last dose of investigational product.
* Participants who, in the opinion of the investigator or the sponsor, will be uncooperative or unable to comply with study procedures.
* Participants who have a newly-diagnosed malignancy or recurrence of malignancy (other than resected cutaneous basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the uterine cervix that has been treated with no evidence of recurrence).
* Participants who have developed any major illness/condition or evidence of an unstable clinical condition (example [e.g.], renal, hepatic, hematologic, gastrointestinal [except disease under study], endocrine, cardiovascular, pulmonary, immunologic [e.g. Felty's syndrome], or local active infection/infectious illness) that, in the investigator's judgment, will substantially increase the risk to the participant if he or she participates in the study.
* Participants with any other severe acute or chronic medical or psychiatric condition or laboratory or ECG abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participants with known exposure to Mycobacterium tuberculosis (TB) since testing at screening in study SHP647-301 (NCT03259334) or SHP647-302 (NCT03259308) and who have been advised to require treatment for latent or active disease, but who are without a generally accepted course of treatment.
* Participants who are investigational site staff members or relatives of those site staff members or participants who are sponsor employees directly involved in the conduct of the study.
* Participants who are participating in other investigational studies (other than SHP647-301, SHP647-302, or SHP647-303) or plan to participate in other investigational studies during long-term extension study SHP647-304.

Participants with Crohn's Disease:

* Participants who had major protocol deviation(s) (as determined by the sponsor) in study SHP647-305, SHP647-306 or SHP647-307.
* Participants who permanently discontinued investigational product because of an adverse events (AE), regardless of relatedness to investigational product, in study SHP647-305, SHP647-306 or SHP647-307.
* Participants who are likely to require major surgery for CD or developed acute severe complications of CD (with or without fulfilling the treatment failure criteria in the maintenance study) that required immediate intervention (e.g. need for immediate biologic treatment with proven effect) and/or Crohn's Disease Activity Index (CDAI) score more than (>) 450.
* Participants are females who became pregnant during study SHP647-305, SHP647-306 or SHP647-307, females who are lactating, females who are planning to become pregnant during the study period, or males or females of childbearing potential not agreeing to continue appropriate contraception methods (i.e. highly effective methods for female and medically appropriate methods for male study participants) through the conclusion of study participation.
* Participants who do not agree to postpone donation of any organ or tissue, including male participants who are planning to bank or donate sperm and female participants who are planning to harvest or donate eggs, for the duration of the study and through 16 weeks after last dose of investigational product.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (417):
- United States (103):
  - Arizona Digestive Health Mesa - East, Mesa, Arizona
  - Elite Clinical Studies - Phoenix - Clinedge - PPDS, Phoenix, Arizona
  - Arizona Digestive Health, Sun City, Arizona
  - CATS Research Center - University of Arizona, Tucson, Arizona
  - Atria Clinical Research - Clinedge - PPDS, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - United Medical Doctors, Encinitas, California
  - University of California San Diego, La Jolla, California
  - OM Research LLC - Lancaster - ClinEdge - PPDS, Lancaster, California
  - Tibor Rubin VA Medical Center - NAVREF, Long Beach, California
  - VA Long Beach Healthcare System - NAVREF - PPDS, Long Beach, California
  - Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - Alliance Clinical Research-(Vestavia Hills), Poway, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of California San Francisco, San Francisco, California
  - Care Access Research, San Pablo, San Pablo, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Asthma and Allergy Associates PC - CRN - PPDS, Colorado Springs, Colorado
  - Renaissance Research Medical Group, INC, Cape Coral, Florida
  - Gastro Florida, Clearwater, Florida
  - Advanced Clinical Research Network, Coral Gables, Florida
  - Alliance Medical Research LLC, Coral Springs, Florida
  - ENCORE Borland-Groover Clinical Research - ERN - PPDS, Jacksonville, Florida
  - SIH Research, Kissimmee, Florida
  - Hi Tech and Global Research, LLc, Miami, Florida
  - Nuren Medical and Research Center, Miami, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - Advanced Clinical Research Network, Miami, Florida
  - Crystal Biomedical Research, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Pharma Research International Inc, Naples, Florida
  - Bayside Clinical Research - New Port Richey, New Port Richey, Florida
  - Omega Research Consultants LLC - Clinedge - PPDS, Orlando, Florida
  - Accel Research Sites - St. Petersburg - ERN - PPDS, Pinellas Park, Florida
  - BRCR Medical Center, Inc, Plantation, Florida
  - East Coast Institute for Research, LLC, Saint Augustine, Florida
  - DBC Research, Tamarac, Florida
  - Gastrointestinal Diseases, Inc Research - IACT- HyperCore - PPDS, Columbus, Georgia
  - Atlanta Center For Gastroenterology PC, Decatur, Georgia
  - Infinite Clinical Trials, Morrow, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Loretto Hospital, Chicago, Illinois
  - IL Gastroenterology Group, Gurnee, Illinois
  - Edward Hines Jr VA Hospital - NAVREF - PPDS, Hines, Illinois
  - Dupage Medical Group, Oakbrook Terrace, Illinois
  - Medisphere Medical Research Center LLC, Evansville, Indiana
  - Laporte County Institute For Clinical Research, Michigan City, Indiana
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Gastroenterology Associates of Hazard, Hazard, Kentucky
  - CroNOLA, LLC., Houma, Louisiana
  - Clinical Trials of SWLA LLC, Lake Charles, Louisiana
  - DelRicht Clinical Research, LLC - ClinEdge - PPDS, New Orleans, Louisiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Commonwealth Clinical Studies LLC, Brockton, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Gastroenterology Associates of Western Michigan, PLC, Wyoming, Michigan
  - Mayo Clinic Health System - PPDS, Duluth, Minnesota
  - Minnesota Gastroenterology PA, Saint Paul, Minnesota
  - Digestive Health Center PA, Ocean Springs, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - St Louis Center For Clinical Research, St Louis, Missouri
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Encompass Care, North Las Vegas, Nevada
  - New York Total Medical Care PC, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Weill Cornell Medical College, New York, New York
  - Southtowns Gastroenterology, PLLC, Orchard Park, New York
  - East Carolina Gastroenterology, Jacksonville, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Gastro Health Research, Cincinnati, Ohio
  - Consultants For Clinical Research Inc, Cincinnati, Ohio
  - Consultants For Clinical Research Inc, Fairfield, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Ohio Clinical Research Partners LLC, Mentor, Ohio
  - Veteran's Research and Education Foundation - NAVREF - PPDS, Oklahoma City, Oklahoma
  - Veterans Research Foundation of Pittsburgh - NAVREF - PPDS, Pittsburgh, Pennsylvania
  - Penn State Hershey Medical Group, State College, Pennsylvania
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Advanced Gastroenterology-Union City, Union City, Tennessee
  - Northside Gastroenterology, Cypress, Texas
  - Digestive Health Associates of Texas, P.A.dba DHAT Research Institute, Garland, Texas
  - Precision Research Institute, LLC, Houston, Texas
  - Biopharma Informatic Inc., Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Aztec Medical Research, Houston, Texas
  - Biopharma Informatic Research Center, Houston, Texas
  - Southern Star Research Institute LLC, San Antonio, Texas
  - DM Clinical Research - ERN - PPDS, Tomball, Texas
  - Inquest Clinical Research/Coastal Gastroenterology Associates, PA - TDDC - PPDS, Webster, Texas
  - HP Clinical Research, Bountiful, Utah
  - Mid Atlantic Health Specialists, Galax, Virginia
  - Winchester Gastroenterology Associates, Winchester, Virginia
  - CHI Franciscan Digestive Care Associates, Tacoma, Washington
  - Exemplar Research, Inc. - Elkins, Elkins, West Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Argentina (3):
  - Fundación Favaloro, Buenos Aires
  - Hospital Privado Centro Médico de Córdoba, Córdoba
  - Sanatorio 9 de Julio SA, San Miguel de Tucumán
- Australia (7):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Box Hill, Victoria
  - St Vincents Hospital Melbourne - PPDS, Melbourne, Victoria
- Austria (7):
  - A.ö. Krankenhaus der Barmherzigen Brüder, Sankt Veit an der Glan, Carinthia
  - LKH-Universitätsklinikum Klinikum Graz, Graz, Styria
  - Klinikum Klagenfurt Am Woerthersee, Klagenfurt
  - Salzburger Landeskliniken, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (4):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven- Gasthuisberg Campus, Leuven, Vlaams Brabant
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - CHU Mouscron, Mouscron
- Clinical Center Banja Luka, Banja Luka, Bosnia and Herzegovina
- Bulgaria (13):
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment EOOD, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment - Dr. Georgi Stranski EAD, Pleven
  - Multiprofile Hospital for Active Treatment Eurohospital, Plovdiv
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases Dr.D.Gramatikov- Ruse- PPDS, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Medical Center Excelsior OOD - PPDS, Sofia
  - Second Multiprofile Hospital for Active Treatment Sofia, Sofia
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sv Ivan Rilski EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna - ISUL EAD, Sofia
  - Medical Center Convex EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment Sveta Anna, Sofia
  - Diagnostic Consultative Centre Mladost - M OOD, Varna
- Canada (2):
  - Percuro Clinical Research LTD, Victoria, British Columbia
  - Toronto Digestive Disease Associates Inc, Toronto, Ontario
- Colombia (4):
  - Hospital Pablo Tobón Uribe, Medellín, Antioquia
  - Servimed S.A.S, Bucaramanga, Santander Department
  - Fundación Valle Del Lili, Cali, Valle del Cauca Department
  - IPS Centro Médico Julián Coronel S.A.S. - PPDS, Cali
- Croatia (8):
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - Opca Bolnica Karlovac, Karlovac, Karlovacka Županija
  - Opca bolnica Bjelovar, Bjelovar
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital Centre Split, Split
  - General Hospital Virovitica, Virovitica
  - General County Hospital Vukovar and Croatian Veterans Hospital, Vukovar
  - General Hospital Zadar, Zadar
- Czechia (6):
  - Hepato-Gastroenterologie HK, s. r. o., Hradec Králové, Královéhradecký kraj
  - PreventaMed s.r.o., Olomouc, Olomoucký kraj
  - Institut Klinicke A Experimentalni Mediciny, Prague
  - ISCARE I.V.F. a.s., Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
  - Nemocnice Pardubickeho kraje, a.s. Orlickoustecka nemocnice, Ústí nad Orlicí
- Estonia (3):
  - OÜ LV Venter, Pärnu, Pärnumaa
  - East Viru Central Hospital, Kohta-Järve
  - West Tallinn Central Hospital, Tallinn
- Germany (12):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum der RWTH Aachen, Aachen, North Rhine-Westphalia
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
  - Gastro Campus Research GbR, Münster, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - Universitatsklinikum Jena, Jena, Thuringia
  - Charité - Universitätsmedizin Berlin, Berlin
  - Gastroenterologische Facharztpraxis am Mexikoplatz, Berlin-Zehlendorf
  - Sana Klinikum Biberach, Biberach an der Riss
  - Universitätsklinikum Frankfurt, Frankfurt
  - Asklepios Westklinikum Hamburg Ggmbh, Hamburg
  - Klinikum rechts der Isa der Technischen Universitaet Muenchen, Munich
- Greece (6):
  - Ippokrateio General Hospital of Athens, Athens, Attica
  - University General Hospital of Heraklion, Heraklion
  - Iatriko Palaiou Falirou, Paliao Faliro
  - University General Hospital of Patras, Pátrai
  - Theageneio Anticancer Oncology Hospital of Thessaloniki, Thessaloniki
  - Euromedica - PPDS, Thessaloniki
- Hungary (12):
  - Bekes Megyei Kozponti Korhaz, Békéscsaba
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
  - ENDOMEDIX Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz, Gyula
  - Mohacsi Korhaz, Mohács
  - Tolna Megyei Balassa János Kórház, Szekszárd
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Jávorszky Ödön Kórház, Vác
  - Csolnoky Ferenc Korhaz, Veszprém
- St Vincent's University Hospital, Dublin, Ireland
- Israel (6):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - PPDS, Jerusalem
  - Galilee Medical Center, Nahariya
  - Nazareth EMMS Hospital, Nazareth
  - Tel Aviv Sourasky Medical Center PPDS, Tel Aviv
  - Baruch Padeh Poriya Medical Center, Tiberias
- Italy (15):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo (FG), Apulia
  - Azienda Ospedaliera Mater Domini Di Catanzaro, Catanzaro, Calabria
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Di Modena Policlinico, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar, Veneto
  - Azienda Ospedale Università Padova, Padua, Veneto
  - A.O.U. Maggiore della Carità, Novara
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - La Sapienza-Università di Roma-Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Japan (35):
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaidô
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Medical Corporation Aoyama Clinic, Kobe, Hyôgo
  - Hyogo College of Medicine, Nishinomiya-shi, Hyôgo
  - Sagamihara Kyodo Hospital, Sagamihara, Kanagawa
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Nihonbashi Egawa Clinic, Chuo-Ku, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Ome Municipal General Hospital, Ōme, Tokyo
  - Tokatsu Tsujinaka Hospital, Abiko
  - Kunimoto Hospital, Asahikawa
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hakodate Koseiin Hakodate Goryoukaku Hospital, Hakodate
  - Yuai Memorial Hospital, Koga
  - Kawabe Clinic, Koganei
  - Hidaka Coloproctology Clinic, Kurume-shi
  - Aizawa Hospital, Matsumoto-shi
  - Aichi Medical University Hospital, Nagakute
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Onomichi General Hospital, Onomichi
  - Chiinkai Dojima General & Gastroenterology Clinic, Osaka
  - Kinshukai Infusion Clinic, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu
  - Bellland General Hospital, Sakai
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Tohoku Rosai Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga-gun
  - Medical Corporation Shoyu-kai Fujita Gastroenterology Hospital, Takatsuki
  - Koukokukai Ebisu Clinic, Tokyo
  - Colo-Proctology Center Matsushima Clinic, Yokohama
  - Shinbeppu Hospital, Beppu, Ôita
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Ôita
  - Yodogawa Christian Hospital, Osaka, Ôsaka
- Lebanon (3):
  - Al Zahraa University Hospital, Beirut
  - Rafik Hariri University Hospital, Beirut
  - Hammoud Hospital University Medical Center, Saida
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santaros Klinikos, Vilnius
  - Vilnius City Clinical Hospital, Vilnius
- Mexico (11):
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Centro de Investigacion Clinica Acelerada, S.C., Tepeyac Insurgentes, Mexico City
  - Clinica de Higado y Gastroenterologia Integral, S.C., Cuernavaca, Morelos
  - JM Research S.C, Cuernavaca, Morelos
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey, Nuevo León
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Centro de Investigación Médica Aguascalientes, Aguascalientes
  - Phylasis Clinicas Research S. de R.L. de C.V., Cuautitlán Izcalli
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Accelerium, S. de R.L. de C.V., Monterrey
  - Clinical Research Institute, Tlalnepantla
- Netherlands (5):
  - ETZ-Elisabeth, Tilburg, North Brabant
  - NWZ, location Alkmaar, Alkmaar, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - VU Medisch Centrum, Amsterdam
  - Amsterdam UMC - Meibergdreef 9, Amsterdam
- New Zealand (4):
  - Auckland City Hospital, Grafton, Auckland
  - Dunedin Hospital, Dunedin, South Island
  - Wellington Hospital, Newtown, Wellington Region
  - Waikato Hospital, Hamilton
- Poland (35):
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o., Włocławek, Kuyavian-Pomeranian Voivodeship
  - Krakowskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - Lexmedica, Wroclaw, Lower Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej CENTRUM MEDYCZNE Szpital Swietej Rodziny, Lódz, Lódzkie
  - Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej Centralny Szpital Weteranow, Lódz, Lódzkie
  - Instytut Centrum Zdrowia Matki Polki, Lódz, Lódzkie
  - BioVirtus Centrum Medyczne, Józefów, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej VIVAMED, Warsaw, Masovian Voivodeship
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok, Podlaskie Voivodeship
  - Endoskopia Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Szpital Zakonu Bonifratrow pw. Aniolow Strozow w Katowicach, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Bydgoszcz- PRATIA - PPDS, Bydgoszcz
  - Centrum Medyczne Czestochowa - PRATIA - PPDS, Częstochowa
  - Centrum Medyczne Gdynia - PRATIA - PPDS, Gdynia
  - NZOZ All Medicus, Katowice
  - Centrum Medyczne A-Z Clinic Mateusz Sidor, Piotr Puc-Lekarze Spolka Partnerska, Krakow
  - Centrum Opieki Zdrowotnej Orkan-Med Stec-Michalska Sp. J., Ksawerów
  - Med Gastr Sp.z.o.o Sp.k, Lodz
  - Twoja Przychodnia NCM, Nowa Sól
  - Centrum Innowacyjnych Terapii, Piaseczno
  - Clinical Research Center Spółka z Ograniczoną Odpowiedzialnością, Medic-R Spółka Komandytowa, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Sonomed Sp. z o.o., Szczecin
  - H-T. Centrum Medyczne Endoterapia, Tychy
  - Centrum Zdrowia MDM, Warsaw
  - Centrum Medyczne Warszawa - PRATIA - PPDS, Warsaw
  - Centralny Szpital Kliniczny MSW, Warsaw
  - Samodzielny Publiczny Szpital Wojewodzki im. Papieza Jana Pawla II, Zamość
  - Szpital Specjalistyczny sw Lukasza - Oddzial Gastroenterologii, Gmina Końskie, Świętokrzyskie Voivodeship
- Portugal (5):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Algarve - Hospital de Portimao, Faro
  - Hospital Senhora da Oliveira - Guimaraes, E.P.E, Guimarães
  - Hospital da Luz, Lisbon
  - Hospital de São Bernardo, Setúbal
- Romania (12):
  - Dr.Carol Davila Emergency University Central Military Hospital, Bucharest
  - Sana Monitoring SRL, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - Fundeni Clinical Institute, Bucharest
  - SC Centrul Medical MEDICUM S.R.L., Bucharest
  - Emergency University Hospital, Bucharest
  - Cluj-Napoca Emergency Clinical County Hospital, Cluj-Napoca
  - Affidea Romania SRL, Constanța
  - Gastromedica SRL, Iași
  - Dr. Tirnaveanu Amelita Private Practice, Oradea
  - Dr. Goldis Gastroenterology Center SRL, Timișoara
- Russia (17):
  - St. Elizabeth Municipal Clinical Hospital, Saint Petersburg, Sankt-Peterburg
  - Kazan State Medical University, Kazan'
  - Moscow Clinical Scientific Center, Moscow
  - Moscow Regional Research Clinical Institute Na Mfvladimirskiy, Moscow
  - Nizhegorodskaya Regional Clinical Hospital n.a. Semashko, Nizhny Novgorod
  - Research Institute of Physiology and Basic Medicine, Novosibirsk
  - Rostov State Medical University, Rostov-on-Don
  - First St. Petersburg State Medical University n.a. I.P Pavlov, Saint Petersburg
  - Union Clinic, LLC, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M. Kirov, Saint Petersburg
  - Medical University Reaviz, Samara
  - Private Healthcare Institution Clinical Hospital RZD-Medicina of Samara city, Samara
  - Medical Company Hepatolog, LLC, Samara
  - SHI Regional Clinical Hospital, Saratov
  - Smolensk Regional Clinical Hospital, Smoensk
  - Stavropol State Medical University, Stavropol
  - Regional Consulting and Diagnostics Centre, Tyumen
- Serbia (5):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - University Clinical Center Nis, Niš
  - General Hospital Vrsac, Vršac
  - Clinical Hospital Center Zemun, Zemun
  - University Clinical Center Kragujevac, Kragujevac, Šumadijski Okrug
- Slovakia (3):
  - Univerzitna nemocnica Bratislava, Bratislava
  - KM Management, spol. s r.o., Nitra
  - Gastro LM, s.r.o., Prešov
- South Africa (3):
  - CLINRESCO, ARWYP Medical Suites, Johannesburg, Gauteng
  - Dr. J Breedt, Pretoria, Gauteng
  - Dr JP Wright, Claremont, Western Cape
- South Korea (14):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang'yeogsi
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gang'weondo
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeonggido
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggido
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center PPDS, Seoul
- Spain (11):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid, Madrid, Communidad Delaware
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Centro Medico Teknon - Grupo Quironsalud, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz - PPDS, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universität Zürich, Zurich, Zürich (de), Switzerland
- Turkey (Türkiye) (2):
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Mersin University Medical Faculty, Mersin
- Ukraine (27):
  - Regional Municipal Non-profit Enterprise "Chernivtsi Regional Clinical Hospital", Chernivtsi, Chernivtsi Oblast
  - Municipal Nonprofit Enterprise CCH #2 n.a. prof. O.O. Shalimov of Kharkiv City Council, Kharkiv, Kharkivs’ka Oblast’
  - Communal Nonprofit Enterprise Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VR, Vinnytsia, Vinnytsia Oblast
  - Municipal Non-profit Enterprise City Emergency Care Hospital of Zaporizhzhia Regional Council, Zaporizhzhia, Zaporizhzhia Oblast
  - ME Dnipropetrovsk Regional Clinical Hospital n.a. I.I Mechnykov Dnipropetrovsk Regional Council, Dnipro
  - LLC Medical Center Family Medicine Clinic, Dnipro
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipro
  - Clinic of SI National Institute of Therapy n.a. L.T. Mala of NAMS of Ukraine, Kharkiv
  - Municipal Nonprofit Enterprise of Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - MNPE of Kharkiv Regional Council Regional Clinical Specialised Dispensary of Radiation Protection, Kharkiv
  - Municipal Non-profit Enterprise Kherson City Clinical Hospital named after Ye.Ye. Karabelesh, Kherson
  - Municipal Enterprise Kryvyi Rih City Clinical Hospital #2 of Kryvyi Rih City Council, Kryvyi Rih
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv
  - Kyiv City Clinical Hospital #18, Kyiv
  - Treatment and Diagnostic Center "Healthy and Happy" of LLC "Healthy and Happy", Kyiv
  - Medical Center OK!Clinic+LLC International Institute of Clinical Research, Kyiv
  - Medical Center of LLC Medical Center Dopomoga-Plus, Kyiv
  - Communal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Hospital, Kyiv
  - Municipal Non-profit Enterprise of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Railway Clinical Hospital of branch Health Center of Joint Stock Co. Ukrainian Railway, Lviv
  - MNE Lviv Territorial Med Ass-n Multidisciplinary Clinical Hospital for Intensive Care and Ambulance, Lviv
  - Municipal Non-profit Enterprise Odessa Regional Clinical Hospital of Odessa Regional Council, Odesa
  - MNPE Central City Clinical Hospital of Uzhhorod City Council, Uzhhorod
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
  - Communal Nonprofit Enterprise Vinnytsia Regional Clinical Hospital named after N.I. Pirogov VRC, Vinnytsia
  - Communal Non-Commercial Enterprise Vinnytsia City Clinical Hospital 1, Vinnytsia
  - MNPE City Hospital No. 6 of Zaporizhzhia City Council, Zaporizhzhia
- United Kingdom (8):
  - Fairfield General Hospital - PPDS, Lancashire, Bury
  - Whipps Cross University Hospital, London, London, City of
  - North Tyneside General Hospital, North Shields, Northumberland
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - Aberdeen Royal Infirmary - PPDS, Aberdeen
  - Western General Hospital Edinburgh - PPDS, Edinburh
  - Royal Gwent Hospital - PPDS, Newport
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe14db2bf003ab476b8

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 225 investigative sites in 33 countries from 27 February 2018 to 13 December 2023.
Pre-assignment Details: Participants from induction and maintenance studies of ulcerative colitis (UC) [SHP647-301 (NCT03259334), SHP647-302 (NCT03259308), and SHP647-303 (NCT03290781)] and Crohn's disease (CD) [SHP647-305 (NCT03559517), SHP647-306 (NCT03566823), and SHP647-307 (NCT03627091)] were enrolled to receive either 25 milligrams (mg) or 75 mg ontamalimab.
Groups:
- UC: Ontamalimab 25 mg: Participants received 25 milligrams (mg) of ontamalimab solution for injection subcutaneously (SC), every 4 weeks (Q4W), for up to 3 years.
- UC: Ontamalimab 25 mg Then 75 mg; CD: Ontamalimab 25 mg Then 75 mg: Participants received 25 mg of ontamalimab solution for injection SC, Q4W, and later progressed to receive 75 mg in a similar manner for up to 5.79 years.
- CD: Ontamalimab 25 mg: Participants received 25 mg of ontamalimab solution for injection SC, Q4W, for up to 3 years.
Period: Overall Study
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Started | 89 | 159 | 268 | 5 | 10 | 26
Completed | 0 | 117 | 129 | 0 | 6 | 12
Not Completed | 89 | 42 | 139 | 5 | 4 | 14
Not completed — Adverse Event | 18 | 3 | 13 | 0 | 0 | 5
Not completed — Death | 0 | 0 | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 42 | 21 | 66 | 3 | 3 | 5
Not completed — Physician Decision | 14 | 8 | 19 | 0 | 0 | 2
Not completed — Site Terminated by Sponsor | 1 | 0 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 12 | 6 | 24 | 1 | 1 | 0
Not completed — Reason not Specified | 0 | 4 | 8 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set included all participants who received at least 1 dose of investigational product (IP) in the SHP647-304 study.
Groups:
- Total: Total of all reporting groups
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg | Total
Number analyzed (Participants) | 89 | 159 | 268 | 5 | 10 | 26 | 557
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 2 | 7 | 0 | 1 | 1 | 11
  Between 18 and 65 years | 87 | 148 | 239 | 4 | 9 | 25 | 512
  >=65 years | 2 | 9 | 22 | 1 | 0 | 0 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 67 | 111 | 1 | 5 | 14 | 227
  Male | 60 | 92 | 157 | 4 | 5 | 12 | 330
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 12 | 15 | 0 | 1 | 2 | 35
  Not Hispanic or Latino | 84 | 146 | 251 | 5 | 9 | 24 | 519
  Unknown or Not Reported | 0 | 1 | 2 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 4 | 0 | 0 | 1 | 7
  Asian | 7 | 14 | 24 | 1 | 0 | 0 | 46
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 4 | 0 | 0 | 2 | 8
  White | 77 | 135 | 231 | 4 | 9 | 23 | 479
  More than one race | 2 | 2 | 3 | 0 | 0 | 0 | 7
  Unknown or Not Reported | 2 | 4 | 2 | 0 | 1 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs (TEAEs) were defined as AEs with start dates or worsening dates at the time of or following the first exposure to investigational product.
Time Frame: From first dose of study drug up to end of study [EOS] (up to 5.79 years)
Population: The Safety Set included all participants who received at least 1 dose of IP in the SHP647-304 study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Number analyzed (Participants) | 89 | 159 | 268 | 5 | 10 | 26
Participants | 67 | 122 | 203 | 4 | 8 | 17

2. Primary Outcome: Number of Participants With Serious Infections
Description: Serious infections were defined as any infections that were life-threatening or those requiring hospitalization or intravenous antibiotics based on the investigator's assessment.
Time Frame: From first dose of study drug up to EOS (up to 5.79 years)
Population: The Safety Set included all participants who received at least 1 dose of IP in the SHP647-304 study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Number analyzed (Participants) | 89 | 159 | 268 | 5 | 10 | 26
Participants | 5 | 4 | 17 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Notable Changes in Clinical Laboratory Parameters Over Time
Description: Clinical laboratory assessments included hematology, serum chemistry and urinalysis. Any notable changes in the clinical laboratory value over time based on the investigator interpretation were reported.
Time Frame: From first dose of study drug up to EOS (up to 5.79 years)
Population: The Safety Set included all participants who received at least 1 dose of IP in the SHP647-304 study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Number analyzed (Participants) | 89 | 159 | 268 | 5 | 10 | 26
Participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Primary Outcome: Number of Participants With Discernible Changes in Electrocardiogram (ECG) Over Time
Description: ECG included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals and corrected QT (QTc) intervals parameters measurement. Any discernible changes in the ECG value over time based on investigator interpretation were reported.
Time Frame: From first dose of study drug up to EOS (up to 5.79 years)
Population: The Safety Set included all participants who received at least 1 dose of IP in the SHP647-304 study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Number analyzed (Participants) | 89 | 159 | 268 | 5 | 10 | 26
Participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

5. Primary Outcome: Number of Participants With Discernible Changes in Vital Signs Over Time
Description: Vital sign assessments included blood pressure, pulse, respiratory rate, and temperature. Any discernible changes in vital signs over time per investigator interpretation were reported.
Time Frame: From first dose of study drug up to EOS (up to 5.79 years)
Population: The Safety Set included all participants who received at least 1 dose of IP in the SHP647-304 study.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Number analyzed (Participants) | 89 | 159 | 268 | 5 | 10 | 26
Participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Number of Participants With Ulcerative Colitis With Treatment Response Over Time
Description: Treatment response over time was defined as clinical composite score that has decreased by greater than or equal to (≥2) points and ≥30 percentage (%), with an accompanying decrease in the sub score for rectal bleeding (RB) ≥1 point or a subscore for RB ≤ 1, and/or composite score that has decreased by ≥30% and ≥3 points compared to the baseline value for induction studies. The clinical composite score is a measure consisting of sub scores RB (0-3) plus stool frequency (0-3) with higher scores indicating more severe disease. With the implementation of amendment 4 of the protocol the study became a single arm study with all participants receiving the 75 mg dose of ontamalimab. Hence, only those UC participants who were receiving the 75 mg dose of ontamalimab every 4 weeks and participating in amendment 4 of the protocol were analyzed in this outcome measure.
Time Frame: Up to 5.79 years
Population: Full Analysis Set (FAS) included all participants in the randomized set who received at least 1 dose of IP in the SHP647-304 study. Overall number analyzed is the number of UC participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | UC: Ontamalimab 25 mg Then 75 mg | UC: Ontamalimab 75 mg
Number analyzed (Participants) | 120 | 133
Participants | 116 | 129

7. Secondary Outcome: Number of Participants With Crohn's Disease With Treatment Response Over Time
Description: Treatment response over time=Crohn's Disease Activity Index(CDAI)score that has decreased ≥100 points and/or simple endoscopic score for Crohn's disease(SES-CD)that has decreased by ≥25%,both compared to baseline value for induction studies.SES-CD is simple scoring system with 4 endoscopic variables measured in same 5 ileocolonic segments as CD index of severity. Overall values on SES-CD range from 0-56,higher values=more severe disease.4 endoscopic variables are scored from 0-3 in each bowel segment:ileum,right/transverse/left colon,rectum. Presence & size of ulcers(none=0;diameter 0.1-0.5centimeter(cm)=1;0.5-2cm=2;>2cm=3);extent of ulcerated surface(none=0;<10%=1;10%-30%=2; >30%= 3);extent of affected surface(none=0;<50%=1;50%-75%=2;>75%=3);Presence & type of narrowing (none=0;single can be passed=1;multiple can be passed=2;cannot be passed=3).
Time Frame: Up to 5.79 years
Population: FAS included all participants in randomized set who received at least 1 dose of IP in the SHP647-304 study. With implementation of protocol amendment 4 this became a single arm study with all participants receiving 75 mg ontamalimab. Hence, only those CD participants who were receiving ontamalimab 75mg Q4W and participating in amendment 4 of the protocol were analyzed. Overall number analyzed is the number of CD participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
Number analyzed (Participants) | 6 | 13
Participants | 6 | 12

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to EOS (up to 5.79 years)
Description: Safety Set included all participants who received at least 1 dose of IP in the SHP647-304 study.
Groups:
- UC: Ontamalimab 25 mg; CD: Ontamalimab 25 mg: Participants received 25 mg of ontamalimab solution for injection SC, Q4W, for up to 3 years.
- UC: Ontamalimab 25mg Then 75 mg: Participants received 25 mg of ontamalimab solution for injection SC, Q4W, and later progressed to receive 75 mg in a similar manner for up to 3 years.Participants received 25 mg of ontamalimab solution for injection SC, Q4W, and later progressed to receive 75 mg in a similar manner for up to 5.79 years.
- UC: Ontamalimab 75mg: Participants received 75 mg of ontamalimab solution for injection SC, Q4W, forup to 5.79 years.
Arm/Group | UC: Ontamalimab 25 mg | UC: Ontamalimab 25mg Then 75 mg | UC: Ontamalimab 75mg | CD: Ontamalimab 25 mg | CD: Ontamalimab 25 mg Then 75 mg | CD: Ontamalimab 75 mg
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/159 | 3/268 | 1/5 | 0/10 | 0/26
Serious Adverse Events (participants affected / at risk) | 15/89 | 21/159 | 46/268 | 2/5 | 2/10 | 4/26
Other Adverse Events (participants affected / at risk) | 47/89 | 109/159 | 155/268 | 3/5 | 8/10 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UC: Ontamalimab 25 mg (N=89) | UC: Ontamalimab 25mg Then 75 mg (N=159) | UC: Ontamalimab 75mg (N=268) | CD: Ontamalimab 25 mg (N=5) | CD: Ontamalimab 25 mg Then 75 mg (N=10) | CD: Ontamalimab 75 mg (N=26)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 1 | 4 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 6 | 3 | 10 | 0 | 0 | 0
Colon dysplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0
Cytomegalovirus gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 1 | 3 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UC: Ontamalimab 25 mg (N=89) | UC: Ontamalimab 25mg Then 75 mg (N=159) | UC: Ontamalimab 75mg (N=268) | CD: Ontamalimab 25 mg (N=5) | CD: Ontamalimab 25 mg Then 75 mg (N=10) | CD: Ontamalimab 75 mg (N=26)
Abdominal pain (Gastrointestinal disorders) | 2 | 11 | 8 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 7 | 14 | 16 | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 3
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 10 | 13 | 0 | 2 | 1
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 10 | 0 | 2 | 1
Blood pressure increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 9 | 8 | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 2 | 3 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 22 | 21 | 28 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 2 | 40 | 57 | 0 | 2 | 4
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 17 | 10 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 3 | 5 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 10 | 9 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 0 | 1 | 0
Eyelid rash (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 8 | 6 | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 16 | 10 | 1 | 1 | 3
Hypertension (Vascular disorders) | 3 | 12 | 13 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 5 | 16 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 8 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 2 | 4 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 18 | 20 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 11 | 5 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 5 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 3 | 2 | 9 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 9 | 13 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 4 | 4 | 0 | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 3 | 4 | 0 | 2 | 0
Rubber sensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 6 | 4 | 0 | 2 | 1
Tongue blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 9 | 16 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03283085/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT03283085/SAP_001.pdf